CLINICAL TRIAL: NCT00382668
Title: Single-Dose Pharmacokinetics of Dasatinib in Subjects With Hepatic Impairment Compared to Healthy Adult Subjects
Brief Title: A Study of Dasatinib to See How Liver Impaired and Healthy Subjects Process and React to the Study Drug
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: CA180-051
Record Dates: First submitted 2006-09-26; First posted 2006-09-29 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Liver Diseases
Keywords: hepatically impaired
MeSH Terms: conditions — Liver Diseases | interventions — Dasatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A
  Interventions: Drug: Dasatinib
- B
  Interventions: Drug: Dasatinib
- C
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 50 mg, once daily, for one day
  Other Names: Sprycel
  Groups: A
Drug: Dasatinib — Tablets, Oral, 20 mg, once daily for one day
  Other Names: Sprycel
  Groups: B
Drug: Dasatinib — Tablets, Oral, 70 mg, once daily for one day
  Other Names: Sprycel
  Groups: C

SUMMARY:
The primary purpose of this study is to evaluate how a person with liver impairment processes and reacts to the study drug. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria - All subjects:

* Male and females ≥18 years old
* Women must be of non-childbearing potential
* Adequate hematologic and renal function
* BMI 18-35 kg/m2

Inclusion Criteria - Liver Impaired subjects:

* Subjects must have stable liver impairment diagnosed with standard classification - Child Pugh

Exclusion Criteria - All subjects:

* Inability to swallow or absorb oral medication
* Uncontrolled medical disorder or infection
* Use of CYP3A4 inhibitors/inducers or drugs with risk of Torsades de Pointes
* Uncontrolled or Significant cardiovascular disease
* Any significant bleeding disorder
* Female subjects of childbearing potential
* Male subjects unwilling to use an effective method of contraception throughout the conduct of the study and for 2 months thereafter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and Female Subjects with hepatic insufficiency conforming to Child-Pugh classification B
  Male and Female Subjects with hepatic insufficiency conforming to Child-Pugh classification C
  Healthy Control subjects in good health
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - University Of Miami, Miami, Florida
  - Comprehensive Phase One, Miramar, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - New Orleans Center For Clinical Research, Knoxville, Tennessee